CLINICAL TRIAL: NCT05870592
Title: Detection of Abnormal Respiratory Cell Populations in Lung Cancer Screening Patients
Brief Title: Detection of Abnormal Respiratory Cell Populations in Lung Cancer Screening Patients Using the CyPath Lung Assay
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: bioAffinity Technologies Inc. (Industry)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Lung Cancer Screening CyPath
Record Dates: First submitted 2023-05-10; First posted 2023-05-23 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are numerous Department of Defense (DoD) beneficiaries enrolled in the various lung cancer screening programs across the DoD. This study may enable patients to forego annual CT lung cancer screening or help to predict cancerous nodules without interventional procedures. This is a prospective observational study of sputum cytology using flow cytometry to analyze sputum samples collected from patients in the active military who are undergoing annual lung cancer screening. The primary objective of this study is to analyze the cellular profiles of sputum samples collected from the Acapella® airway assist device in patients at higher risk for lung cancer. The target population are high risk patients for developing lung cancer, age 50-80 with a significant smoking history.

DETAILED DESCRIPTION:
There are numerous Department of Defense (DoD) beneficiaries enrolled in the various lung cancer screening programs across the DoD. This is a prospective observational study of sputum cytology using flow cytometry to analyze sputum samples collected from patients undergoing annual lung cancer screening. The primary objective of this study is to analyze the cellular profiles of sputum samples collected with the assistance of the Acapella® airway assist device in patients at higher risk for lung cancer. The target population are high risk patients for developing lung cancer, age 50-80 with a significant smoking history.

A sputum sample will be collected by the patient over a three-day period at home using the Acapella® airway assist device (Smiths Medical). The Acapella device is a noninvasive airway resistance device to assist with coughing to clear airway mucous in patients with bronchiectasis and other similar disorders. Male and female participants who are in the active military and who are at high risk for lung cancer and undergoing an annual low dose CT (LDCT) of the chest to assess for new nodules will be enrolled. Individuals at high risk for lung cancer include participants who are 50-80 years of age, have smoked the equivalent of one pack of cigarettes a day for 30 years or more, and who have not quit smoking in the past 15 years. Patients will be selected on the presence or absence of new CT findings; half of the cohort will have no new CT findings and the other half of the cohort will have new changes on CT suggestive of possible malignancy.

Participants who sign an informed consent and satisfy the inclusion/exclusion criteria will be enrolled into the research study. The sputum sample will be collected by the participant at home over a three (3) day period (1 sample/day) using the Acapella© airway assist device in accordance with device instructions. Subjects will pool their 3 sputum samples into one collection cup and return the cup to the collection site at the Brooke Army Medical Center Pulmonary Clinic within 2 weeks after completing their scheduled LDCT. Participants will use the Acapella® to loosen their mucus and aid in the collection of the sputum sample. The study coordinator will instruct the participant at Visit 1 in the use of the Acapella® in accordance with device instructions. After use of the acapella®, the participant will be instructed to wait five minutes for mucus to collect at the back of the throat and then start to huff cough to expel sputum. The participant will then be instructed to spit sputum without scraping their throat by coughing into the sample collection cup. Participants should receive a collection cup, the Acapella® device, and instructions to take home. Participants should collect all three samples in the single collection cup over three days at home. After the third sputum collection at home using the Acapella®, the participant will return the combined sputum sample in one collection cup to the collection site.

Upon receipt by the collection site, sputum samples will be refrigerated and shipped the same day, if possible, with a cold pack to the bioAffinity (BA) laboratory for processing using the CyPath Lung Assay. Acquisition of data on cells in the sputum samples will be done by BA researchers using the Navios flow cytometer at Precision Pathology Services (PPS).

Sputum samples will be collected in a sterile collection cup without preservative and kept refrigerated (2-8 °C) until shipping. Patients will keep their specimens refrigerated until delivered to the Pulmonary Clinic. Samples will be kept refrigerated in the Pulmonary Clinic until shipping. At the BA laboratories, the sample will be processed, labeled with antibodies and dyes to identify cell populations, and thereafter data will be acquired and analyzed by flow cytometry. Sample processing will be performed under a safety hood. Sputum sample preparation for flow cytometry analysis consists of chemical dissociation of sputum to produce a single cell suspension sample that is labeled with fluorescently labeled antibodies that distinguishes leukocyte populations such as granulocytes, alveolar macrophages, and T and B lymphocytes. Antibodies also specifically stain non-inflammatory cell types such as squamous epithelial cells in the sputum. The sputum sample is labeled with the fluorescent porphyrin meso-tetra-(4-carboxyphenyl) (TCPP) that preferentially binds to cancer cells and cancer-related cells in sputum. A viability stain is used to eliminate dead cells from the analysis, including contaminating squamous epithelial cells (cheek cells). The gating strategy also excludes doublets and debris from analysis. The presence of alveolar macrophages confirms the sample is from the airways.

Specimens collected by the collection site will not be labeled with subject identification other than uniquely assigned study participant numbers. The individual responsible for accessioning the samples will not be the same person performing any of the assays. Consequently, BA researchers will be blinded as to the identity of the participants.

Researchers blinded to the participant's identity will perform the experiments that compare the characteristics of samples. Findings from this research will not be given to providers to diagnose malignancy in participants or utilized in subsequent treatment decisions.

If the sample collection is inadequate, patients will be given a single additional collection kit to resubmit the sputum sample.

The following clinical data will be collected for each patient.

1. Demographics (age, gender, height, weight)
2. Medical and surgical history to include pulmonary diseases.
3. Medication use
4. Smoking history
5. Results from the most recent low dose CT (LDCT) for the presence/absence of new findings.

ELIGIBILITY:
Inclusion Criteria:

* Active Military
* 50-80 years-of-age
* Smoking history of 20-pack-years or more
* If not currently smoking cigarettes, quit smoking within 15 years of giving sputum sample
* Undergoing CT scan of chest as part of annual screening for lung cancer

Exclusion Criteria:

* Active respiratory illness in the preceding 2 weeks
* Using antibiotics in the past 2 weeks
* Unable to use Acapella device for sputum collection
* Known history of lung cancer

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from the BAMC Pulmonary lung cancer screening tracker. After completion fo their annual LDCT, patients will be asked if they wish to participate in the study and provide a 3-day sputum sample. If they request to participate, they will meet with one of the study investigators to provide written informed consent. Once consented, they will be provided with an Acapella device and instructed on the use for sample collection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 12 months
  The primary objective of this study is to analyze the cellular profiles of sputum samples collected from the Acapella® airway assist device in patients at higher risk for lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Morris, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Hospital, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grayson M, Lai SC, Bederka LH, Araujo P, Sanchez J, Reveles XT, Rebel VI, Rebeles J. Quality-Controlled Sputum Analysis by Flow Cytometry. J Vis Exp. 2021 Aug 9;(174). doi: 10.3791/62785. PMID 34424239
- [Background] Bederka LH, Sanchez JR, Rebeles J, Araujo PR, Grayson MH, Lai SC, DePalo LR, Habib SA, Hill DG, Lopez K, Patriquin L, Sussman R, Humphreys J, Reveles XT, Rebel VI. Sputum analysis by flow cytometry; an effective platform to analyze the lung environment. PLoS One. 2022 Aug 17;17(8):e0272069. doi: 10.1371/journal.pone.0272069. eCollection 2022. PMID 35976857
- [Background] Elzi DJ, Bauta WE, Sanchez JR, Das T, Mogare S, Zannes Fatland P, Iza M, Pertsemlidis A, Rebel VI. Identification of a novel mechanism for meso-tetra (4-carboxyphenyl) porphyrin (TCPP) uptake in cancer cells. FASEB J. 2021 Mar;35(3):e21427. doi: 10.1096/fj.202000197R. PMID 33629776
- [Result] Lemieux ME, Reveles XT, Rebeles J, Bederka LH, Araujo PR, Sanchez JR, Grayson M, Lai SC, DePalo LR, Habib SA, Hill DG, Lopez K, Patriquin L, Sussman R, Joyce RP, Rebel VI. Detection of early-stage lung cancer in sputum using automated flow cytometry and machine learning. Respir Res. 2023 Jan 21;24(1):23. doi: 10.1186/s12931-023-02327-3. PMID 36681813
- [Result] Patriquin L, Merrick DT, Hill D, Holcomb RG, Lemieux ME, Bennett G, Karia B, Rebel VI, Bauer T 2nd. Early Detection of Lung Cancer with Meso Tetra (4-Carboxyphenyl) Porphyrin-Labeled Sputum. J Thorac Oncol. 2015 Sep;10(9):1311-1318. doi: 10.1097/JTO.0000000000000627. PMID 26200451